CLINICAL TRIAL: NCT00138671
Title: Efficacy and Safety of Inhaled Human Insulin (Exubera) Compared With Subcutaneous Human Insulin in the Therapy of Adult Subjects With Type 1 or Type 2 Diabetes Mellitus and Chronic Obstructive Pulmonary Disease: A One-Year, Multicenter, Randomized, Outpatient, Open-Label, Parallel-Group Comparative Trial
Brief Title: A One Year Clinical Trial Assessing the Usefulness and Safety of Inhaled Insulin in Diabetics With COPD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171030
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitus; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous Insulin (Active Comparator)
  Interventions: Drug: Subcutaneous Insulin
- Inhaled Insulin (Experimental)
  Interventions: Drug: Inhaled Insulin

INTERVENTIONS:
Drug: Subcutaneous Insulin — Subcutaneous short-acting insulin with dose adjusted according to premeal blood glucose plus oral antidiabetic agent(s) and/or either once or twice daily doses of either Ultralente or neutral protamine hagedorn (NPH) insulin, or a single bedtime dose of insulin glargine.
  Arms: Subcutaneous Insulin
Drug: Inhaled Insulin — Inhaled insulin with dose adjusted according to premeal blood glucose plus oral antidiabetic agent(s) and/or either once or twice daily doses of either Ultralente or NPH insulin, or a single bedtime dose of insulin glargine.
  Arms: Inhaled Insulin

SUMMARY:
A One Year Clinical Trial Assessing the Usefulness and Safety of Inhaled Insulin in Diabetics with Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing Exubera. At that time recruitment for study A2171030 was placed on hold. Nektar, the company from which Pfizer licensed Exubera, announced on April 9, 2008 that it had stopped its search for a new marketing partner. Accordingly, there will be no commercial availability of Exubera. As a result, study A2171030 was terminated on June 17, 2008. Neither safety nor efficacy reasons were the cause of the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus (Type 1 or Type 2) currently controlled with injected insulin
* Prior smokers with a fixed airflow obstruction at screening (FEV1/FVC < 70%) and FEV1 < 80% predicted and/or a history of chronic productive cough.

Exclusion Criteria:

* Poorly controlled, unstable or steroid-dependent COPD, insulin pump therapy, active smoking

Ages: 30 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2003-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (62):
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Searcy, Arkansas
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Lake City, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Honululu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Normal, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Waltham, Massachusetts
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Fredericksburg, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Huntington, West Virginia
  - Pfizer Investigational Site, Madison, Wisconsin
- Brazil (3):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (5):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site, San José, Provincia de San José, Costa Rica
- Pfizer Investigational Site, Neuss, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171030&StudyName=A%20One%20Year%20Clinical%20Trial%20Assessing%20the%20Usefulness%20and%20Safety%20of%20Inhaled%20Insulin%20in%20Diabetics%20with%20COPD

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Insulin: Inhaled insulin with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin: Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Period: Overall Study
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Started | 59 | 46
Completed | 46 | 30
Not Completed | 13 | 16
Not completed — Death | 0 | 3
Not completed — Adverse Event | 6 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Insulin | Subcutaneous Insulin | Total
Number analyzed (Participants) | 59 | 46 | 105
Age, Customized [Number; unit: participants]
  36 to 45 years | 1 | 3 | 4
  46 to 55 years | 10 | 4 | 14
  56 to 65 years | 20 | 23 | 43
  66 to 75 years | 27 | 15 | 42
  > 75 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 42 | 37 | 79
Primary Diagnosis (Diabetes Type I or II) [Number; unit: participants] — Type I or Type II diabetes mellitus was defined using the American Diabetes Association criteria (2002).
  participants
    Type I | 7 | 6 | 13
    Type II | 52 | 40 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was measured in liters (L) 30 minutes following the administration of ipratropium. Change from baseline: mean of (value of observed FEV1 (L) at treatment duration minus baseline value).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 12, 18, 26, 39, 52
Population: Full Analysis Set (FAS), FEV1=all randomized subjects who received at least 1 dose of study treatment, had a baseline FEV1 measurement (post-bronchodilator), and had at least 1 FEV1 post-baseline measurement (post-bronchodilator). Number of subjects with evaluable data: n=Inhaled Insulin, Subcutaneous Insulin.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 59 | 43
L
  Week 1 (n=52, 39) | -0.021 (0.132) | -0.018 (0.125)
  Week 2 (n=51, 40) | -0.039 (0.116) | -0.042 (0.120)
  Week 3 (n=47, 40) | -0.026 (0.121) | -0.048 (0.145)
  Week 4 (n=50, 38) | -0.050 (0.140) | -0.039 (0.151)
  Week 6 (n=53, 38) | -0.045 (0.152) | -0.070 (0.165)
  Week 12 (n=48, 41) | -0.056 (0.180) | -0.007 (0.187)
  Week 18 (n=52, 37) | -0.049 (0.158) | -0.071 (0.195)
  Week 26 (n=52, 38) | -0.067 (0.174) | -0.096 (0.189)
  Week 39, (n=47, 34) | -0.053 (0.174) | -0.092 (0.232)
  Week 52 (n=45, 30) | -0.068 (0.208) | -0.128 (0.184)

2. Secondary Outcome: Full Pulmonary Function Tests (PFTs) (Spirometry, Pre-Ipratropium and Pre-Insulin PFTs)
Description: Full PFTs included spirometry pre- and 30-minutes post-ipratropium and were completed between the hours of 6 AM and 10 AM with subjects in the fasting state. Full PFT data were collected, but not analyzed.
Time Frame: Duration of the study
Measure: Number; unit: L
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Full PFTs (DLco, Pre-Ipratropium and Pre- Insulin PFTs)
Description: Full PFTs included DLco pre- and 30-minutes post-ipratropium and were completed between the hours of 6 AM and 10 AM with subjects in the fasting state. Full PFT data were collected, but not analyzed.
Time Frame: Duration of the study
Measure: Number; unit: mL/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change From Baseline in Post-Bronchodilator Carbon Monoxide Diffusion Capacity (DLco)
Description: DLco measured in milliters/minutes/millimeters of mercury (mL/min/mmHg) 30 minutes following the administration of ipratropium. Change from baseline: mean of (value of observed DLco (mL/min/mmHg) at treatment duration minus baseline value).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 12, 18, 26, 39, 52
Population: FAS, FEV1=all randomized subjects who received at least 1 dose of study treatment, had a baseline FEV1 measurement (post-bronchodilator), and had at least 1 FEV1 post-baseline measurement (post-bronchodilator). Number of subjects with evaluable data: n=Inhaled Insulin, Subcutaneous Insulin.
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 59 | 43
mL/min/mmHg
  Week 1 (n=51, 40) | -0.263 (1.610) | -0.319 (0.984)
  Week 2 (n=51, 40) | -0.491 (1.288) | -0.031 (1.106)
  Week 3 (n=47, 40) | -0.494 (1.175) | 0.169 (1.303)
  Week 4 (n=50, 39) | -0.640 (1.345) | -0.482 (1.321)
  Week 6 (n=52, 38) | -0.625 (1.356) | -0.576 (1.226)
  Week 12 (n=47, 40) | -0.379 (1.516) | -0.534 (1.506)
  Week 18 (n=51, 36) | -0.287 (1.463) | -0.286 (1.796)
  Week 26 (n=52, 38) | -0.287 (1.841) | -0.947 (1.643)
  Week 39 (n=47, 33) | -0.611 (1.475) | -0.891 (2.137)
  Week 52 (n=45, 29) | -0.614 (1.754) | -0.882 (1.720)

5. Secondary Outcome: Other PFTs (Besides FEV1 and DLco)
Description: Other PFTs (besides FEV1 and DLco) were measured 30 minutes following the administration of ipratropium. Other PFTs included forced vital capacity (FVC), peak expiratory flow rate (maximal forced expiratory flow) (PEFR[FEFmax]), and forced expiratory flow from 25% to 75% of vital capacity (FEF25%-75%). Other PFT data were collected, but not analyzed.
Time Frame: Duration of the study
Measure: Number; unit: mL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Bronchodilator Responsiveness as Determined by the Change in FEV1
Description: Responsiveness was the percent change from the FEV1 value before bronchodilator use to the FEV1 value 30 minutes after bronchodilator use, operationally defined as [(post-bronchodilator FEV1 minus pre-bronchodilator FEV1 divided by pre-bronchodilator FEV1] multiplied by 100.
Time Frame: Weeks 1, 2, 3, 4, 6, 12, 18, 26, 39, 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 59 | 43
percent change
  Week 1 (n=52, 39) | 4.890 (5.727) | 5.693 (7.249)
  Week 2 (n=51, 40) | 6.132 (6.200) | 5.245 (6.254)
  Week 3 (n=47, 40) | 6.346 (7.469) | 5.820 (8.347)
  Week 4 (n=50, 38) | 5.177 (7.211) | 6.382 (9.685)
  Week 6 (n=53, 38) | 5.988 (6.034) | 7.736 (10.139)
  Week 12 (n=48, 41) | 6.473 (8.994) | 5.542 (6.791)
  Week 18 (n=52, 37) | 6.700 (6.020) | 5.152 (8.155)
  Week 26 (n=52, 38) | 5.585 (5.592) | 5.856 (8.562)
  Week 39 (n=47, 34) | 6.634 (5.829) | 6.098 (9.311)
  Week 52 (n=45, 30) | 6.030 (4.700) | 5.445 (8.390)

7. Secondary Outcome: Insulin Dose Responsiveness for FEV1
Description: FEV1 dose responsiveness 10 and 60 minutes after insulin. FEV1 dose-responsiveness to insulin (defined as the difference between the FEV1 value following a dose of insulin and FEV1 value before a dose of insulin, operationally defined as the post-dose FEV1 value minus pre-dose FEV1 value).
Time Frame: Baseline, Week 9, Week 51
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 50 | 39
L
  Baseline, 10 minutes (n=50, 39) | 0.009 (0.076) | 0.022 (0.106)
  Baseline, 60 minutes (n=50, 39) | -0.004 (0.096) | 0.020 (0.127)
  Week 9, 10 minutes (n=42, 31) | -0.004 (0.110) | 0.016 (0.096)
  Week 9, 60 minutes (n=42, 30) | 0.011 (0.109) | 0.030 (0.116)
  Week 51, 10 minutes (n=46, 31) | -0.021 (0.121) | -0.002 (0.084)
  Week 51, 60 minutes (n=45, 31) | 0.005 (0.115) | -0.020 (0.141)

8. Secondary Outcome: Insulin Dose Responsiveness for DLco
Description: DLco dose responsivness 10 and 60 minutes after insulin. DLco dose-responsiveness to insulin (defined as the difference between the DLco value following a dose of insulin and DLco value before a dose of insulin, operationally defined as the post-dose DLco value minus pre-dose DLco value).
Time Frame: Baseline, Week 9, Week 51
Population: FAS, FEV1=all randomized subjects who received at least 1 dose of study treatment, had a baseline FEV1 measurement (post-bronchodilator), and had a FEV1 post-baseline measurement (post-bronchodilator). Number of subjects with evaluable data: n=Inhaled Insulin, Subcutaneous Insulin.
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 48 | 39
mL/min/mmHg
  Baseline, 10 minutes (n=48, 39) | -0.461 (1.157) | -0.195 (0.707)
  Baseline, 60 minutes (n=49, 39) | -0.597 (1.102) | -0.160 (1.217)
  Week 9, 10 minutes (n=41, 30) | -0.182 (1.015) | -0.238 (1.505)
  Week 9, 60 minutes (n=42, 29) | 0.013 (2.288) | -0.373 (1.574)
  Week 51, 10 minutes (n=44, 31) | -0.465 (0.781) | 0.054 (1.204)
  Week 51, 60 minutes (n=44, 31) | -0.395 (0.885) | -0.163 (1.211)

9. Secondary Outcome: Methacholine PC20
Description: Methacholine challenge testing was conducted at selected sites at visits which did not occur at other sites (Weeks -2.9, -0.9, 11, 50 and 52+5). Methacholine challenge was not analyzed as there was only 1 test performed, which was a baseline test, and no methacholine tests performed in subjects using inhaled insulin.
Time Frame: Duration of the study
Measure: Number; unit: mg/mL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mean Weekly Number of Puffs of Short-Acting Bronchodilator Used
Description: All subjects used diary cards to record their daily use of short-acting bronchodilators. Subjects recorded the sum of their short-acting bronchodilator use (puffs of albuterol plus ipratropium plus Combivent®, as applicable) daily, immediately upon arising, and again in the evening or before bed. Mean weekly number of puffs of short-acting bronchodilator used data were collected, but not analyzed.
Time Frame: Duration of the study
Measure: Number; unit: puffs
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incidence of Non-Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Non-severe COPD exacerbation = additional therapy (systemic corticosteroids, antibiotics, oxygen) needed for worsening respiratory symptoms and/or lung function, not needing hospitalization > 24 hours. Crude event rate = total events divided by subject-months. Subject-months=elapsed number of months a subject was in the study in each time interval.
Time Frame: 0 to 1 week to > 9 months
Population: as for outcome 4
Measure: Number; unit: events/subject-month (crude event rate)
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 59 | 43
events/subject-month (crude event rate)
  0 to 1 week (n=59, 43) | 0.00 | 0.00
  > 1 to 2 weeks (n=59, 43) | 0.07 | 0.00
  > 2 to 3 weeks (n=59, 43) | 0.00 | 0.00
  > 3 to 4 weeks (n=59, 42) | 0.07 | 0.10
  > 4 to 6 weeks (n=57, 42) | 0.08 | 0.05
  > 6 to 9 weeks (n=56, 42) | 0.05 | 0.03
  > 9 to 12 weeks (n=55, 41) | 0.05 | 0.07
  > 3 to 6 months (n=52, 41) | 0.02 | 0.01
  > 6 to 9 months (n=52, 37) | 0.01 | 0.01
  > 9 months (n=50, 35) | 0.01 | 0.02
  Overall (n=59, 43) | 0.02 | 0.02

12. Secondary Outcome: Incidence of Severe COPD Exacerbations
Description: Severe COPD exacerbation = a COPD-related hospitalization > 24 hours. Crude event rate = total events divided by subject-months. Subject-months=elapsed number of months a subject was in the study in each time interval.
Time Frame: 0 to 1 week to > 9 months
Population: as for outcome 4
Measure: Number; unit: events/subject-month (crude event rate)
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 59 | 43
events/subject-month (crude event rate)
  0 to 1 week (n=59, 43) | 0.00 | 0.00
  > 1 to 2 weeks (n=59, 43) | 0.00 | 0.00
  > 2 to 3 weeks (n=59, 43) | 0.00 | 0.00
  > 3 to 4 weeks (n=59, 42) | 0.00 | 0.00
  > 4 to 6 weeks (n=57, 42) | 0.00 | 0.00
  > 6 to 9 weeks (n=56, 42) | 0.00 | 0.00
  > 9 to 12 weeks (n=55, 41) | 0.00 | 0.00
  > 3 to 6 months (n=52, 41) | 0.00 | 0.00
  > 6 to 9 months (n=52, 37) | 0.01 | 0.00
  > 9 months (n=50, 35) | 0.00 | 0.00
  Overall (n= 59, 43) | 0.00 | 0.00

13. Secondary Outcome: Baseline Dyspnea Index (BDI) and Transition Dyspnea Index (TDI) Questionnaires
Description: The BDI and TDI measured or quantitated the severity of breathlessness (shortness of breath) in symptomatic subjects. BDI and TDI data were collected, but not analyzed.
Time Frame: Duration of the study
Measure: Number; unit: grade
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Change from baseline: mean of (value of observed HbA1c at treatment duration minus baseline value).
Time Frame: Baseline, Weeks 6, 12, 26, 39, and 52
Population: FAS, HbA1c=all randomized subjects who received at least 1 dose of study treatment, had a baseline HbA1c measurement, and had at least 1 HbA1c post-baseline measurement. Week 52 Last Observation Carried Forward (LOCF)=subjects' last measurement carried forward. Number of subjects with evaluable data: n=Inhaled Insulin, Subcutaneous Insulin.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 57 | 43
percent
  Week 6 (n=56, 40) | -0.40 (0.81) | -0.48 (0.60)
  Week 12 (n=50, 41) | -0.53 (0.98) | -0.42 (0.65)
  Week 26 (n=52, 38) | -0.39 (0.96) | -0.32 (0.79)
  Week 39 (n=48, 35) | -0.34 (1.11) | -0.20 (1.01)
  Week 52 (n=46, 32) | -0.30 (1.10) | -0.23 (0.84)
  Week 52 LOCF (n=57, 43) | -0.28 (1.03) | -0.26 (0.79)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.10, 90% CI [-0.17 to 0.36]
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.01, 90% CI [-0.27 to 0.26]
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Test type: Superiority or Other; Mean Difference (Final Values) = -0.02, 90% CI [-0.29 to 0.26]
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Test type: Superiority or Other; Mean Difference (Final Values) = -0.08, 90% CI [-0.36 to 0.20]
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 90% CI [-0.23 to 0.35]
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 LOCF; Test type: Superiority or Other; Mean Difference (Final Values) = 0.01, 90% CI [-0.29 to 0.31]

15. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Change from baseline: mean of (value of observed fasting plasma glucose in milligrams/deciliters (mg/dL) at treatment duration minus baseline value).
Time Frame: Baseline, Weeks 6, 12, 26, 39, 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 57 | 43
mg/dL
  Week 6 (n=52, 39) | -24.67 (69.69) | 2.89 (41.17)
  Week 12 (n=48, 39) | -30.73 (52.99) | -0.18 (46.25)
  Week 26 (n=47, 38) | -34.92 (61.63) | 10.45 (62.80)
  Week 39 (n=47, 33) | -20.45 (56.62) | 10.43 (98.53)
  Week 52 (n=45, 31) | -23.40 (65.77) | 12.37 (58.01)
  Week 52 (LOCF) (n=57, 43) | -28.55 (65.85) | 2.36 (66.51)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Test type: Superiority or Other; Mean Difference (Final Values) = -4.475, 90% CI [-23.47 to 14.518]
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -10.91, 90% CI [-30.04 to 8.232]
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Test type: Superiority or Other; Mean Difference (Final Values) = -22.84, 90% CI [-42.51 to -3.166]
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Test type: Superiority or Other; Mean Difference (Final Values) = -8.222, 90% CI [-28.52 to 12.075]
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Test type: Superiority or Other; Mean Difference (Final Values) = -8.329, 90% CI [-29.27 to 12.616]
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 LOCF; Test type: Superiority or Other; Mean Difference (Final Values) = 1.406, 90% CI [-13.70 to 16.514]

16. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline: mean of (value of observed body weight in kilograms (kg) at treatment duration minus baseline value).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 9, 11, 12, 18, 26, 39, 50, 51, 52
Population: FAS, HbA1c=randomized subjects with >=1 study drug dose, baseline and >=1 post-baseline HbA1c measurement. Last Observation Carried Forward (LOCF) method used. Number of subjects with evaluable data: n=Inhaled Insulin, Subcutaneous Insulin. Week 11 and 50 visits were part of the methacholine substudy and were not required visits for all subjects.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 59 | 43
kg
  Week 1 (n=52, 40) | 0.25 (1.62) | 0.02 (0.98)
  Week 2 (n=51, 40) | 0.26 (1.77) | 0.15 (1.73)
  Week 3 (n=49, 41) | 0.19 (2.03) | 0.13 (1.90)
  Week 4 (n=53, 41) | 0.19 (1.98) | 0.24 (2.13)
  Week 6 (n=54, 39) | 0.42 (2.26) | 0.26 (1.94)
  Week 9 (n=47, 34) | 0.31 (2.93) | 0.25 (2.31)
  Week 11 (n=8, 8) | 0.03 (2.25) | -0.14 (2.97)
  Week 12 (n=49, 41) | 0.42 (3.29) | 0.34 (3.69)
  Week 18 (n=52, 37) | 0.40 (3.66) | 0.90 (4.01)
  Week 26 (n=52, 38) | 0.85 (3.95) | 1.99 (4.03)
  Week 39 (n=47, 34) | 0.61 (4.37) | 2.43 (5.21)
  Week 50 (n=8, 6) | 1.75 (4.90) | 6.33 (9.06)
  Week 51 (n=23, 17) | 1.21 (4.82) | 2.67 (3.28)
  Week 52 (n=43, 27) | 0.97 (5.65) | 3.32 (4.68)
  Week 52 LOCF (n=59, 43) | 0.99 (4.20) | 2.40 (4.79)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 1; Test type: Superiority or Other; Mean Difference (Final Values) = 0.884, 90% CI [-0.317 to 2.084]
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 2; Test type: Superiority or Other; Mean Difference (Final Values) = 0.470, 90% CI [-0.728 to 1.668]
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 3; Test type: Superiority or Other; Mean Difference (Final Values) = 0.382, 90% CI [-0.815 to 1.579]
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 4; Test type: Superiority or Other; Mean Difference (Final Values) = 0.405, 90% CI [-0.793 to 1.602]
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Test type: Superiority or Other; Mean Difference (Final Values) = 0.562, 90% CI [-0.642 to 1.766]
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 9; Test type: Superiority or Other; Mean Difference (Final Values) = 0.416, 90% CI [-0.809 to 1.641]
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 11; Test type: Superiority or Other; Mean Difference (Final Values) = 0.019, 90% CI [-1.416 to 1.454]
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.091, 90% CI [-1.127 to 1.308]
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 18; Test type: Superiority or Other; Mean Difference (Final Values) = -0.309, 90% CI [-1.551 to 0.934]
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Test type: Superiority or Other; Mean Difference (Final Values) = -0.869, 90% CI [-2.123 to 0.384]
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Test type: Superiority or Other; Mean Difference (Final Values) = -1.664, 90% CI [-2.968 to -0.360]
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 50; Test type: Superiority or Other; Mean Difference (Final Values) = -2.116, 90% CI [-3.829 to -0.403]
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 51; Test type: Superiority or Other; Mean Difference (Final Values) = -1.801, 90% CI [-3.204 to -0.397]
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Test type: Superiority or Other; Mean Difference (Final Values) = -2.026, 90% CI [-3.384 to -0.668]
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 LOCF; Test type: Superiority or Other; Mean Difference (Final Values) = -1.451, 90% CI [-3.003 to 0.101]

17. Secondary Outcome: Mean Total Daily Intermediate-/Long-Acting Insulin Dose (Unadjusted for Body Weight)
Description: Intermediate-/long-acting insulin included Insulin NPH, Ultralente, and Insulin Glargine for both groups.
Time Frame: Weeks 1, 2, 3, 4, 6, 9, 12, 18, 26, 39, 52
Population: FAS, HbA1c=all randomized subjects who received at least 1 dose of study treatment, had a baseline HbA1c measurement, and had at least 1 HbA1c post-baseline measurement. Number of subjects with evaluable data: n=Inhaled Insulin, Subcutaneous Insulin.
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 51 | 43
Units
  Week 1 (n=53, 40) | 43.78 (22.20) | 48.18 (23.44)
  Week 2 (n=50, 41) | 44.96 (22.50) | 48.04 (24.33)
  Week 3 (n=51, 39) | 47.04 (24.36) | 50.53 (24.44)
  Week 4 (n=52, 41) | 47.50 (25.94) | 50.30 (25.61)
  Week 6 (n=54, 40) | 49.56 (26.61) | 51.34 (25.91)
  Week 9 (n=47, 35) | 48.68 (28.61) | 56.72 (25.89)
  Week 12 (n=51, 41) | 49.23 (28.46) | 52.32 (29.49)
  Week 18 (n=51, 40) | 50.87 (29.32) | 53.83 (29.34)
  Week 26 (n=51, 38) | 50.47 (28.83) | 55.78 (28.11)
  Week 39 (n=49, 35) | 49.99 (29.00) | 53.10 (26.11)
  Week 52 (n=48, 34) | 50.66 (30.63) | 53.39 (26.32)

18. Secondary Outcome: Mean Total Daily Short-Acting Insulin Dose (Unadjusted for Body Weight)
Description: Short-acting insulin (mg) for the Inhaled Insulin group was Inhaled Insulin. Short-acting insulin (unit) for the Subcutaneous Insulin group included Insulin Lispro, Insulin Aspart, and Regular Insulin.
Time Frame: Weeks 1, 2, 3, 4, 6, 9, 12, 18, 26, 39, 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mg, Units
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 56 | 41
mg, Units
  Week 1 (n=54, 40) | 12.34 (5.26) | 32.74 (21.59)
  Week 2 (n=51, 41) | 13.03 (6.63) | 32.08 (22.25)
  Week 3 (n=52, 39) | 14.10 (6.89) | 32.88 (21.60)
  Week 4 (n=53, 41) | 14.17 (7.28) | 31.85 (22.29)
  Week 6 (n=55, 40) | 15.17 (7.20) | 33.42 (22.72)
  Week 9 (n=48, 35) | 15.82 (7.41) | 36.65 (22.94)
  Week 12 (n=52, 41) | 15.64 (7.80) | 33.58 (23.94)
  Week 18 (n=52, 40) | 16.47 (7.48) | 35.36 (26.06)
  Week 26 (n=52, 38) | 16.71 (8.05) | 37.73 (26.14)
  Week 39 (n=49, 35) | 17.22 (8.60) | 37.47 (26.20)
  Week 52 (n=48, 34) | 16.85 (9.52) | 39.28 (25.13)

19. Secondary Outcome: Mean Total Daily Intermediate-/Long-Acting Insulin Dose (Adjusted for Body Weight)
Description: Intermediate/long-acting insulin included Insulin NPH, Ultralente, and Insulin Glargine for both groups. Dose was adjusted for body weight (units divided by kg).
Time Frame: Weeks 1, 2, 3, 4, 6, 9, 12, 18, 26, 39, 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units/kg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 51 | 43
Units/kg
  Week 1 (n=51, 40) | 0.46 (0.22) | 0.48 (0.19)
  Week 2 (n=50, 40) | 0.47 (0.22) | 0.48 (0.20)
  Week 3 (n=49, 39) | 0.50 (0.25) | 0.50 (0.21)
  Week 4 (n=50, 41) | 0.49 (0.26) | 0.50 (0.21)
  Week 6 (n=53, 39) | 0.52 (0.27) | 0.51 (0.21)
  Week 9 (n=46, 34) | 0.50 (0.29) | 0.57 (0.21)
  Week 12 (n=49, 41) | 0.51 (0.28) | 0.52 (0.24)
  Week 18 (n=51, 37) | 0.53 (0.29) | 0.55 (0.24)
  Week 26 (n=51, 38) | 0.52 (0.28) | 0.55 (0.22)
  Week 39 (n=47, 34) | 0.51 (0.27) | 0.54 (0.24)
  Week 52, (n=43, 27) | 0.52 (0.29) | 0.56 (0.21)

20. Secondary Outcome: Mean Total Daily Short-Acting Insulin Dose (Adjusted for Body Weight)
Description: Short-acting insulin (mg) for the Inhaled Insulin group was Inhaled Insulin. Short-acting insulin (unit) for the Subcutaneous Insulin group included Insulin Lispro, Insulin Aspart, and Regular Insulin. Dose was adjusted for body weight (mg divided by kg or units divided by kg).
Time Frame: Weeks 1, 2, 3, 4, 6, 9, 12, 18, 26, 39, 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mg/kg, Units/kg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 56 | 41
mg/kg, Units/kg
  Week 1 (n=52, 40) | 0.13 (0.05) | 0.33 (0.21)
  Week 2 (n=51, 40) | 0.14 (0.06) | 0.33 (0.21)
  Week 3 (n=49, 39) | 0.15 (0.07) | 0.33 (0.22)
  Week 4 (n=51, 41) | 0.15 (0.07) | 0.32 (0.22)
  Week 6 (n=54, 39) | 0.16 (0.07) | 0.34 (0.22)
  Week 9 (n=47, 34) | 0.17 (0.07) | 0.36 (0.22)
  Week 12 (n=49, 41) | 0.17 (0.08) | 0.34 (0.23)
  Week 18 (n=52, 37) | 0.17 (0.08) | 0.37 (0.24)
  Week 26 (n=52, 38) | 0.18 (0.08) | 0.38 (0.24)
  Week 39 (n=47, 34) | 0.18 (0.08) | 0.38 (0.25)
  Week 52 (n=43, 27) | 0.18 (0.09) | 0.40 (0.25)

21. Secondary Outcome: Lipids
Description: Lipids collected: Total cholesterol, high-density lipoprotein, low-density lipoptrotein, and triglycerides. Lipids data were collected, but not analyzed.
Time Frame: Duration of the study
Measure: Number; unit: mg/dL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Hypoglycemic Event Rates
Description: A hypoglycemic event was identified by characteristic symptoms; blood glucose levels at 59 mg/dL (3.2 mmol/L) or less with a glucose check; or any glucose measurement 49 mg/dL (2.7 mmol/L) or less, with or without symptoms. Crude event rate=total events divided by subject-months. Subject-months=elapsed number of months a subject was in the study in each time interval.
Time Frame: 0 to1 month to > 11 months
Population: as for outcome 17
Measure: Number; unit: events / subject-month
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 57 | 43
events / subject-month
  0 to 1 month (n=57, 43) | 1.76 | 1.36
  > 1 to 2 months (n=56, 42) | 1.25 | 0.98
  > 2 to 3 months (n=55, 42) | 1.21 | 0.97
  > 3 to 4 months (n=52, 41) | 0.87 | 0.67
  > 4 to 5 months (n=52, 40) | 0.96 | 1.01
  > 5 to 6 months (n=52, 38) | 0.69 | 1.13
  > 6 to 7 months (n=52, 37) | 0.62 | 0.92
  > 7 to 8 months (n=51, 36) | 0.67 | 0.75
  > 8 to 9 months (n=51, 36) | 0.59 | 0.78
  > 9 to 10 months (n=51, 36) | 0.50 | 0.52
  > 10 to 11 months (n=49, 34) | 0.75 | 0.51
  > 11 months (n=47, 33) | 0.62 | 0.26
  Overall (n=57, 43) | 0.89 | 0.84

23. Secondary Outcome: Severe Hypoglcyemic Event Rates
Description: An event was severe if the subject was unable to treat him/herself; had at least 1 neurological symptom; or blood glucose of < = 49 mg/dL or the blood glucose was not measured, but the clinical manifestations were reversed by oral carbohydrates, subcutaneous glucagon, or intravenous glucose. Crude event rate=total events/100 subject-months. Subject-months=elapsed number of months a subject was in the study in each time interval.
Time Frame: 0 to 1 month to > 11 months
Population: as for outcome 17
Measure: Number; unit: events / 100 subject-months
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 57 | 43
events / 100 subject-months
  0 to 1 month (n=57, 43) | 1.71 | 2.35
  > 1 to 2 months (n=56, 42) | 1.79 | 0.00
  > 2 to 3 months (n=55, 42) | 0.00 | 0.00
  > 3 to 4 months (n=52, 41) | 0.00 | 0.00
  > 4 to 5 months (n=52, 40) | 0.00 | 0.00
  > 5 to 6 months (n=52, 38) | 0.00 | 0.00
  > 6 to 7 months (n=52, 37) | 0.00 | 0.00
  > 7 to 8 months (n=51, 36) | 0.00 | 0.00
  > 8 to 9 months (n=51, 36) | 1.96 | 0.00
  > 9 to 10 months (n=51, 36) | 2.01 | 0.00
  > 10 to 11 months (n=49, 34) | 0.00 | 0.00
  > 11 months (n=47, 33) | 0.00 | 0.00
  Overall (n=57, 43) | 0.64 | 0.22

ADVERSE EVENTS:
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Serious Adverse Events (participants affected / at risk) | 17 | 14
Other Adverse Events (participants affected / at risk) | 59 | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Inhaled Insulin | Subcutaneous Insulin
Anaemia (Blood and lymphatic system disorders) | 1/59 | 0/46
Angina unstable (Cardiac disorders) | 1/59 | 0/46
Coronary artery disease (Cardiac disorders) | 0/59 | 2/46
Myocardial infarction (Cardiac disorders) | 1/59 | 3/46
Inguinal hernia (Gastrointestinal disorders) | 0/59 | 1/46
Intestinal obstruction (Gastrointestinal disorders) | 0/59 | 1/46
Nausea (Gastrointestinal disorders) | 0/59 | 1/46
Vomiting projectile (Gastrointestinal disorders) | 0/59 | 1/46
Chest pain (General disorders) | 1/59 | 0/46
Hypothermia (General disorders) | 0/59 | 1/46
Ill-defined disorder (General disorders) | 0/59 | 1/46
Implant site erosion (General disorders) | 1/59 | 0/46
Appendicitis (Infections and infestations) | 0/59 | 1/46
Cellulitis (Infections and infestations) | 1/59 | 0/46
Gastroenteritis viral (Infections and infestations) | 0/59 | 1/46
Osteomyelitis (Infections and infestations) | 0/59 | 1/46
Pneumonia (Infections and infestations) | 3/59 | 0/46
Postoperative wound infection (Infections and infestations) | 1/59 | 0/46
Drug administration error (Injury, poisoning and procedural complications) | 0/59 | 1/46
Radius fracture (Injury, poisoning and procedural complications) | 1/59 | 0/46
Rib fracture (Injury, poisoning and procedural complications) | 1/59 | 0/46
Wrist fracture (Injury, poisoning and procedural complications) | 1/59 | 0/46
Electrocardiogram abnormal (Investigations) | 0/59 | 1/46
Troponin increased (Investigations) | 0/59 | 1/46
Dehydration (Metabolism and nutrition disorders) | 1/59 | 0/46
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/59 | 0/46
Hypoglycaemia (Metabolism and nutrition disorders) | 1/59 | 1/46
Ketoacidosis (Metabolism and nutrition disorders) | 1/59 | 0/46
Back pain (Musculoskeletal and connective tissue disorders) | 0/59 | 1/46
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/59 | 0/46
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/59 | 0/46
Depressed level of consciousness (Nervous system disorders) | 1/59 | 0/46
Neuropathy peripheral (Nervous system disorders) | 1/59 | 0/46
Syncope (Nervous system disorders) | 0/59 | 1/46
Azotaemia (Renal and urinary disorders) | 0/59 | 1/46
Bladder neck obstruction (Renal and urinary disorders) | 0/59 | 1/46
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2/59 | 0/46
Arteriosclerosis (Vascular disorders) | 1/59 | 0/46
Hypertension (Vascular disorders) | 0/59 | 1/46
Hypotension (Vascular disorders) | 1/59 | 0/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Inhaled Insulin | Subcutaneous Insulin
Anaemia (Blood and lymphatic system disorders) | 4/59 | 1/46
Coronary artery disease (Cardiac disorders) | 2/59 | 3/46
Myocardial infarction (Cardiac disorders) | 1/59 | 3/46
Vision blurred (Eye disorders) | 2/59 | 4/46
Constipation (Gastrointestinal disorders) | 3/59 | 0/46
Diarrhoea (Gastrointestinal disorders) | 4/59 | 3/46
Nausea (Gastrointestinal disorders) | 4/59 | 4/46
Toothache (Gastrointestinal disorders) | 3/59 | 1/46
Vomiting (Gastrointestinal disorders) | 3/59 | 3/46
Asthenia (General disorders) | 9/59 | 5/46
Chest pain (General disorders) | 4/59 | 1/46
Fatigue (General disorders) | 6/59 | 3/46
Oedema peripheral (General disorders) | 5/59 | 6/46
Seasonal allergy (Immune system disorders) | 3/59 | 0/46
Bronchitis (Infections and infestations) | 8/59 | 2/46
Gastroenteritis (Infections and infestations) | 3/59 | 0/46
Gastroenteritis viral (Infections and infestations) | 2/59 | 3/46
Influenza (Infections and infestations) | 4/59 | 2/46
Nasopharyngitis (Infections and infestations) | 10/59 | 6/46
Otitis media (Infections and infestations) | 3/59 | 1/46
Pneumonia (Infections and infestations) | 4/59 | 2/46
Sinusitis (Infections and infestations) | 3/59 | 2/46
Upper respiratory tract infection (Infections and infestations) | 12/59 | 6/46
Urinary tract infection (Infections and infestations) | 4/59 | 1/46
Contusion (Injury, poisoning and procedural complications) | 3/59 | 2/46
Hypoglycaemia (Metabolism and nutrition disorders) | 40/59 | 30/46
Arthralgia (Musculoskeletal and connective tissue disorders) | 7/59 | 2/46
Back pain (Musculoskeletal and connective tissue disorders) | 5/59 | 5/46
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/59 | 5/46
Myalgia (Musculoskeletal and connective tissue disorders) | 0/59 | 3/46
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/59 | 3/46
Dizziness (Nervous system disorders) | 8/59 | 7/46
Headache (Nervous system disorders) | 10/59 | 3/46
Neuropathy peripheral (Nervous system disorders) | 4/59 | 3/46
Tremor (Nervous system disorders) | 4/59 | 5/46
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4/59 | 4/46
Cough (Respiratory, thoracic and mediastinal disorders) | 5/59 | 2/46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6/59 | 2/46
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3/59 | 0/46
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3/59 | 1/46
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7/59 | 9/46
Hypertension (Vascular disorders) | 6/59 | 3/46

LIMITATIONS AND CAVEATS:
This study was terminated due to Pfizer's decision to stop marketing Exubera®. Due to inconsistency in concomitant medication data entry, interpretation of the event rates for non-severe exacerbations may be of limited clinical value.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.